CLINICAL TRIAL: NCT06172985
Title: A CCTA Image Assisted Triage Software for the Assessment of Patients With Suspected Coronary Artery Disease: a Retrospective, Multi-center, Blind-evaluation Study
Brief Title: A CCTA Image Assisted Triage Software for the Assessment of Patients With Suspected Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Keya Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-091-2022
Record Dates: First submitted 2023-08-17; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-08

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected patients with coronary heart disease.: The coronary CT angiography (CCTA) images collected by each center within a certain period of time will be desensitized after the screening is successful. The final CCTA images were sent to an independent judgment expert group for diagnosis, the results of the test group and the independent judgment expert group were compared, and the clinical application of the coronary artery CT angiography image vascular stenosis auxiliary triage software developed by Keya Medical Technology Co., Ltd. was evaluated. Validity and Accuracy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Due to observational study

SUMMARY:
The goal of this clinical trail is to evaluate the effectiveness and accuracy of the CCTA image assisted triage software(DeepVessel® Cardisight, Keya Medical.) for the triage of patients with suspected coronary artery disease.

DETAILED DESCRIPTION:
The CCTA images collected by each center within a certain period of time would be screened, desensitized, and then evaluated by the software and independent expert group respectively, to evaluate the effectiveness and accuracy of the coronary CT angiography image stenosis assisted triage software developed by Koyal Medical Technology Co.

Experiment group: Evaluated by the software Independent expert group: Evaluated by experts (≥5 years of CCTA experience required)

ELIGIBILITY:
Inclusion Criteria:

1. CCTA images acquired by CT detectors need to meet the following requirements:

   * Check Modal = CT
   * Number of detector rows ≥ 64 rows
   * Layer thickness ≤1mm
   * Layer spacing ≤1mm
   * Pixel pitch ≤ 0.5mm
   * Ball tube voltage ≥ 70kV
   * Number of layers ≥ 100 layers
2. CCTA image quality score ≥ 3 (5-point Likert scale).

Exclusion Criteria:

1. Severe coronary artery calcification, which in the judgment of readers affects the stenosis adjudicator;
2. Previous percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG);
3. Congenital anomalies of coronary artery origin or other malformations;
4. Coronary artery occlusive lesions;
5. Implantation of the pacemaker, internal defibrillator electrode, or prosthetic heart valve.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Suspected patients with coronary heart disease.
Sampling Method: Probability Sample
Enrollment: 1093 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of experiment group in triage for patients with suspected coronary artery disease | October 13,2022 to March 1,2023
  Based on the results of the independent expert group, uses stenosis degree≥50% as the boundary for triage indication on a per-patient basis.

SECONDARY OUTCOMES:
Diagnostic time | October 13,2022 to March 1,2023
  Independent expert group: recording the sum of image post-processing time (T1) and the time to produce the results (T2); Experimental group: recording the time from image post-processing to outputting results; Calculate the difference between the two groups.
Patient as research unit | October 13,2022 to March 1,2023
  Evaluation criteria were established based on the results of the independent expert group to evaluate the total conformity rate, KAPPA value, positive predictive value (PPV) and negative predictive value (NPV) of triage tips for patients with suspected coronary heart disease in the experimental group.
Blood vessels were used as the research unit | October 13,2022 to March 1,2023
  Evaluation criteria were established based on the results of the independent expert group to evaluate the total conformity rate, KAPPA value, positive predictive value (PPV) and negative predictive value (NPV) of triage tips for patients with suspected coronary heart disease in the experimental group.
The vascular segment was used as the research unit | October 13,2022 to March 1,2023
  Evaluation criteria were established based on the results of the independent expert group to evaluate the total conformity rate, KAPPA value, positive predictive value (PPV) and negative predictive value (NPV) of triage tips for patients with suspected coronary heart disease in the experimental group.
Gender stratified statistics, respectively, with patients and blood vessels as research units | October 13,2022 to March 1,2023
  Evaluation criteria were established based on the results of the independent expert group to evaluate the sensitivity and specificity of the trial group to the triage hints of suspected patients with coronary heart disease
Manufacturer stratified statistics, respectively, with patients and blood vessels as research units | October 13,2022 to March 1,2023
  Evaluation criteria were established based on the results of the independent expert group to evaluate the sensitivity and specificity of the trial group to the triage hints of suspected patients with coronary heart disease
Row number stratified statistics, respectively, with patients and blood vessels as research units | October 13,2022 to March 1,2023
  Evaluation criteria were established based on the results of the independent expert group to evaluate the sensitivity and specificity of the trial group to the triage hints of suspected patients with coronary heart disease
The stratified statistics of tube voltage were conducted with patients and blood vessels as research units | October 13,2022 to March 1,2023
  Evaluation criteria were established based on the results of the independent expert group to evaluate the sensitivity and specificity of the trial group to the triage hints of suspected patients with coronary heart disease
Layer thickness stratified statistics, patients and blood vessels were used as research units | October 13,2022 to March 1,2023
  Evaluation criteria were established based on the results of the independent expert group to evaluate the sensitivity and specificity of the trial group to the triage hints of suspected patients with coronary heart disease
The patients and blood vessels were selected as the research units | October 13,2022 to March 1,2023
  Evaluation criteria were established based on the results of the independent expert group to evaluate the sensitivity and specificity of the trial group to the triage hints of suspected patients with coronary heart disease
Post-processing image quality evaluation | October 13,2022 to March 1,2023
  Calculate the percentage of post-processing images with the image quality score of 2 or above in the total post-processing images, and the difference between the independent expert group and experimental group.
Software performance evaluation | October 13,2022 to March 1,2023
  From the function of use, ease of operation, stability to evaluate, divided into satisfactory, general, unsatisfactory three levels.

OTHER OUTCOMES:
Device Defects | October 13,2022 to March 1,2023
  In the course of clinical trials, there are unreasonable risks that may endanger human health and life safety under normal use of medical devices, such as label errors, quality problems, and frequent failures

CONTACTS AND LOCATIONS:
Overall Officials: Bin Lu, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (5):
- China (5):
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The Pearl River Hospital of Southern Medical University, Guangzhou, Guangdong
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The First Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Huanggang Central Hospital, Huanggang, Hubei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meijboom WB, Meijs MF, Schuijf JD, Cramer MJ, Mollet NR, van Mieghem CA, Nieman K, van Werkhoven JM, Pundziute G, Weustink AC, de Vos AM, Pugliese F, Rensing B, Jukema JW, Bax JJ, Prokop M, Doevendans PA, Hunink MG, Krestin GP, de Feyter PJ. Diagnostic accuracy of 64-slice computed tomography coronary angiography: a prospective, multicenter, multivendor study. J Am Coll Cardiol. 2008 Dec 16;52(25):2135-44. doi: 10.1016/j.jacc.2008.08.058. PMID 19095130
- [Result] Lucke C, Foldyna B, Andres C, Boehmer-Lasthaus S, Grothoff M, Nitzsche S, Gutberlet M, Lehmkuhl L. Post-processing in cardiovascular computed tomography: performance of a client server solution versus a stand-alone solution. Rofo. 2014 Dec;186(12):1111-21. doi: 10.1055/s-0034-1366726. Epub 2014 Aug 14. PMID 25122171
- [Result] Choi AD, Marques H, Kumar V, Griffin WF, Rahban H, Karlsberg RP, Zeman RK, Katz RJ, Earls JP. CT Evaluation by Artificial Intelligence for Atherosclerosis, Stenosis and Vascular Morphology (CLARIFY): A Multi-center, international study. J Cardiovasc Comput Tomogr. 2021 Nov-Dec;15(6):470-476. doi: 10.1016/j.jcct.2021.05.004. Epub 2021 Jun 12. PMID 34127407
- [Result] Paul JF, Rohnean A, Giroussens H, Pressat-Laffouilhere T, Wong T. Evaluation of a deep learning model on coronary CT angiography for automatic stenosis detection. Diagn Interv Imaging. 2022 Jun;103(6):316-323. doi: 10.1016/j.diii.2022.01.004. Epub 2022 Jan 26. PMID 35090845
- [Result] Meyer M, Schoepf UJ, Fink C, Goldenberg R, Apfaltrer P, Gruettner J, Vajcs D, Schoenberg SO, Henzler T. Diagnostic performance evaluation of a computer-aided simple triage system for coronary CT angiography in patients with intermediate risk for acute coronary syndrome. Acad Radiol. 2013 Aug;20(8):980-6. doi: 10.1016/j.acra.2013.02.014. Epub 2013 Jun 2. PMID 23735619
- [Derived] Chen Y, Yu H, Fan B, Wang Y, Wen Z, Hou Z, Yu J, Wang H, Tang Z, Li N, Jiang P, Wang Y, Yin W, Lu B. Diagnostic performance of deep learning-based coronary computed tomography angiography in detecting coronary artery stenosis. Int J Cardiovasc Imaging. 2025 May;41(5):979-989. doi: 10.1007/s10554-025-03383-0. Epub 2025 Mar 29. PMID 40156689
- See also: Guerbet. Xenetix® 350: Comparative Assessment of Image Quality for Coronary CT Angiography (X-ACT)[EB/OL] — http://www.clinicaltrials.gov/ct2/show/NCT01255722?term=NCT01255722&draw=2&rank=1